CLINICAL TRIAL: NCT06914752
Title: TENS for Endometriosis Pain in Adolescents and Young Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Boskey, Co-Director of Research, Division of Gynecology, Boston Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00050840
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis (Diagnosis)
Keywords: endometriosis; TENS; transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Endometriosis; Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Delayed intervention trial. Individuals will be randomized to immediate or delayed treatment with the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Immediate intervention (Experimental)
  Interventions: Device: TENS
- Delayed Intervention (Experimental)
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — transcutaneous electrical nerve stimulation

SUMMARY:
The goal of this project is plan to investigate the utility of Transcutaneous Electrical Nerve Stimulators (TENS) for the reduction of pain and the improvement of quality of life in adolescents and young adults with chronic pelvic pain related to endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls and young women (13-25)
* Diagnosis of endometriosis,
* Current pelvic pain (score ≥ 3 on Visual Analog Scale, where 0 represents absence of pain and 10 indicates unbearable pain) present for ≥ 14 days/month over the 2 months prior to study enrollment.
* Personal smart phone or mobile device
* Speak either English or Spanish.

Ages: 10 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain - Visual Acuity Scale | 6 months
  Pain on a scale of 0-10, where a higher score indicates worse pain.

SECONDARY OUTCOMES:
Endometriosis Health Profile 30 (EHP-30) | 6 months
  The Endometriosis Health Profile is a 30 item patient-reported outcome measures designed to assess the health-related quality of life of people living with endometriosis. Scores range from 0 to 100 with higher scores being associated with WORSE health related quality of life.
Missed school/work | 6 months
  Individuals will be asked to track the number of days of missed school/work.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No